CLINICAL TRIAL: NCT04563221
Title: Prostatic Artery Embolization (PAE) Using LC Bead LUMI for the Treatment of Symptomatic Benign Prostatic Hyperplasia (BPH)
Brief Title: Prostatic Artery Embolization for the Treatment of Symptomatic Benign Prostatic Hyperplasia (BPH)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding not approved
Sponsor: Andrew Picel (Other)
Responsible Party: Sponsor-Investigator, Andrew Picel, Assistant Clinical Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 51982
Record Dates: First submitted 2020-09-20; First posted 2020-09-24 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Benign Prostatic Hyperplasia; Lower Urinary Tract Symptoms
Keywords: Benign prostatic hyperplasia (BPH); Prostatic artery embolization (PAE); Lower urinary tract symptoms (LUTS); Prostate artery embolization
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Balloon occlusion microcatheter (Experimental): Participants will undergo the PAE procedure using LC Bead LUMI delivered through a balloon occlusion microcatheter.
  Interventions: Device: Prostatic artery embolization
- Standard microcatheter (Experimental): Participants will undergo the PAE procedure using LC Bead LUMI delivered through a standard microcatheter.
  Interventions: Device: Prostatic artery embolization

INTERVENTIONS:
Device: Prostatic artery embolization — Prostatic artery embolization is performed using LC Bead LUMI, which is the investigational device. The particles are administered to the prostatic arteries using either a balloon occlusion or standard microcatheter. Follow-up is performed at 1 month, 6 months, 12 months, and 24 months after intervention.

SUMMARY:
This is a single center, prospective, investigational study to evaluate the safety and efficacy of prostatic artery embolization (PAE) for the treatment of moderate to severe lower urinary tract symptoms (LUTS) due to benign prostatic hyperplasia (BPH). Embolization will be performed with LC Bead LUMI particles using a balloon occlusion microcatheter or standard microcatheter.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 45 years and ≤ 85 years old
* Prostate volume ≥ 40 mL and ≤ 300 mL
* Diagnosis of BPH with moderate to severe lower urinary tract symptoms (LUTS)
* Refractory or intolerant to medical management
* Ineligibility for or refusal of surgical management
* No evidence of prostate cancer

Exclusion Criteria:

* History of pelvic cancer
* Neurogenic bladder disorder
* Bladder diverticula greater than 5 cm or bladder stones
* Acute urinary retention with Foley catheter dependence
* Active urinary tract infection, interstitial cystitis, or prostatitis within the last 3 months
* Prior surgical prostate intervention
* Active participation in another clinical trial

Ages: 45 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with treatment related adverse events assessed by CTCAE v4.0. | 12 months post PAE
Mean change from baseline in symptom score using the IPSS scale at 6 months | Baseline and 6 months post PAE

SECONDARY OUTCOMES:
Mean change from baseline in Qmax (maximum urinary flow) | Baseline, 6 months and 12 months post PAE
Mean change from baseline in PVR (post void residual) | Baseline, 6 months and 12 months post PAE
Mean change from baseline in prostate volume | Baseline, 6 months and 12 months post PAE
Mean change from baseline in IPSS to measure long-terms subjective outcome | Baseline, 12 and 24 months post PAE

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Picel, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No